CLINICAL TRIAL: NCT03874858
Title: A Phase II, Single-arm Study of De-escalation and Treatment-free Remission in Patients With Chronic Myeloid Leukemia Treated With Nilotinib in First-line Therapy Followed by a Second Attempt After Nilotinib and Asciminib Combination: DANTE Study
Brief Title: A Study of Full Treatment-free Remission in Patients With Chronic Myeloid Leukemia
Acronym: DANTE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107AIT15; 2024-516122-66-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2019-03-05; First posted 2019-03-14 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Chronic Myeloid Leukemia (CML); Chronic Myeloid Leukemia - Chronic Phase (CML-CP); Deep Molecular Response (DMR); sustained deep molecular response (sustained DMR); Treatment-Free Remission (TFR); Treatment-Free Remission failure (TFR failure); Full Treatment-Free Remission (FTFR); Tyrosine Kinase Inhibitor (TKI); quantitative Polymerase Chain Reaction (qPCR); digital droplet Polymerase Chain Reaction (ddPCR); ABL001 (Asciminib); AMN107 (Nilotinib); Tasigna; adult
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase | interventions — nilotinib; asciminib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TFR1 stage- Nilotinib (Experimental): During TFR1 stage, all patients will be treated with nilotinib 300 mg QD for up to 48 weeks (consolidation period).
  * Patients with sustained DMR at the end of the consolidation period will enter the TFR1 period and nilotinib will be discontinued.
  * Patients with loss of MMR will return to the standard nilotinib administration
  * Patients with ≥ MMR, but without sustained DMR at the end of the consolidation period will be treated with nilotinib 300 mg QD
  Interventions: Drug: Nilotinib
- TFR2 stage- Nilotinib+Asciminib (Experimental): During the TFR2 stage, participants will be treated with nilotinib and asciminib for up to 96 weeks (reinduction period).
  * Patients with sustained DMR at the end of reinduction will enter TFR2 and asciminib + nilotinib will be discontinued.
  * Patients with ≥ MMR, but without sustained DMR, at the end of the reinduction, will be treated with nilotinib monotherapy at 300 mg BID until the end of the TFR2 stage.
  * Patients with loss of MMR at any time during reinduction or during nilotinib monotherapy will be discontinued from the study.
  Interventions: Drug: Nilotinib; Drug: Asciminib

INTERVENTIONS:
Drug: Nilotinib — Nilotinib oral 300 mg QD hard capsules
  Other Names: AMN107
  Arms: TFR1 stage- Nilotinib
Drug: Nilotinib — Nilotinib oral 300 mg BID hard capsules
  Other Names: AMN107
  Arms: TFR2 stage- Nilotinib+Asciminib
Drug: Asciminib — Asciminib orally at a dose of 40 mg BID film-coated tablets (FCT)
  Other Names: ABL001
  Arms: TFR2 stage- Nilotinib+Asciminib

SUMMARY:
This study is constituted of two stage: Treatment-Free Remission 1 (TFR1) stage and Treatment-Free Remission 2 (TFR2) stage.

The purpose of the TFR1 stage is to assess the effect of nilotinib reduced to half the standard dose for 12 months on treatment-free remission in patients with Chronic Myeloid Leukemia - Chronic Phase (CML-CP) treated with first-line nilotinib who reached a sustained deep molecular response before entering the study.

The purpose of the TFR2 stage is to evaluate whether the use of asciminib in combination with nilotinib after failure of a first attempt at TFR can lead to higher and more durable TFR rates after a second attempt at TKI discontinuation than those reported in other studies.

DETAILED DESCRIPTION:
This is a prospective, single arm, phase II study constituted of two stage: Treatment-Free Remission 1 (TFR1) stage and Treatment-Free Remission 2 (TFR2) stage.

The TFR1 stage is made up of 4 periods:

1. Screening (week -4 - week 0)
2. Nilotinib consolidation (week 0 - week 48): Patients will be treated with nilotinib 300 mg QD. At the end or during the consolidation period, patients will proceed as follows:

   * Patients with sustained DMR at the end of the consolidation phase will enter the treatment-free remission (TFR1) and nilotinib will be discontinued. If two or more consecutive quarterly BCR-ABL RQ-PCR assessments are not performed or results are not available, the patient will not be eligible for TFR1 period and will be treated with nilotinib 300 mg QD until the end of the TFR1 stage (week 144).
   * Patients with loss of major molecular response (MMR) at any time during the consolidation phase will enter the follow-up period and will return to the standard nilotinib administration regimen (nilotinib 300 mg BID) until the end of the TFR1 stage (week 144).
   * Patients with more than MMR, but without meeting the definition of sustained DMR, will remain in the consolidation phase and will be treated with nilotinib 300 mg QD until the end of the TFR1 stage (week 144).
3. Nilotinib treatment-free remission (TFR1) (week 48 - week 144): During the TFR1 period, BCR-ABL levels will be monitored until the end of the TFR1 stage (week 144)
4. Follow up: Patients who remain on half-dose nilotinib after week 48 and patients with loss of MMR at any time during the study will enter follow-up until week 144.

Patients discontinued from the treatment for any reason will be followed for survival information until week 144. All patients still on study treatment at the end of the study will be transitioned to prescription nilotinib.

The TFR2 stage will include two cohorts; an internal cohort made up of patients who participated in the TFR1 stage of this study, and an external cohort of patients who failed a first attempt at TFR with nilotinib outside of this study. The TFR2 stage is made up of 4 periods:

1. Screening for reinduction
2. Reinduction (week 0-96): Patients will be treated with asciminib 40 mg BID + nilotinib 300 mg BID for 96 weeks. Patients will proceed as follows:

   * Patients with sustained DMR at the end of reinduction will enter TFR2 and asciminib + nilotinib will be discontinued. If two or more consecutive quarterly BCR-ABL RQ-PCR assessments are not performed or results are not available, the patient will not be eligible for TFR2
   * Patients not eligible for TFR2 but with more than an MMR continue treatment with asciminib + nilotinib until the end of reinduction (week 96) and then continue nilotinib monotherapy at 300 mg BID until the end of the TFR2 stage (week 144).
   * Patients with loss of MMR at any time during reinduction or during nilotinib monotherapy will be discontinued from the study.
3. Asciminib+nilotinib treatment-free remission (TFR2) (week 96-week 144): During the TFR2 period, BCR-ABL levels will be monitored every month for one year
4. Follow up: Patients with loss of MMR during TFR2 and patients not eligible for TFR2 but with more than an MMR will be treated with nilotinib 300 mg BID and monitored until week 144. If MMR loss occurs during reinduction or during nilotinib monotherapy, patients will be discontinued from the study and treated according to clinical practice.

ELIGIBILITY:
Inclusion Criteria TFR1 stage:

1. Male and female patients 18 years or older.
2. Diagnosis of CML-CP according to the World Health Organization (WHO).
3. Patients with CML-CP under first-line treatment with nilotinib at the approved daily dose of 300 mg BID mg for at least 3 calendar years.

   Note: At study entry, an ongoing treatment at a dose ≥400 mg per day is allowed.
4. Sustained DMR defined as ≥ MR 4.0 (BCR-ABL level ≤0.01% IS) in all of the last 4 BCR-ABL RQ-PCR assessments with a minimum interval between each assessment of 3 months and a maximum interval of 6 months.
5. Patient must meet the following laboratory values at the screening visit:

   * Absolute Neutrophil Count ≥1.0 x 109/L
   * Platelets ≥75 x 109/L
   * Hemoglobin (Hgb) ≥ 9 g/dL
   * Serum creatinine < 1.5 mg/dL
   * Aspartate transaminase (AST) ≤ 3.0 x ULN
   * Alanine transaminase (ALT) ≤ 3.0 x ULN
   * Serum lipase ≤ 2 x ULN
6. Eastern Cooperative Oncology Group performance status (ECOG) 0-2.
7. Study subjects must be able to comply with study procedures and follow-up examinations.
8. Signed informed consent to the TFR1 stage from the patient or from his/her legal representative.

Exclusion Criteria TFR1 stage:

1. Patients with known atypical transcript.
2. CML treatment resistant mutation(s) (T315I, E255K/V, Y253H, F359C/V) detected if testing was done in the past (there is no requirement to perform mutation testing at study entry if it was not done in the past).
3. Dose reductions/interruptions due to neutropenia or thrombocytopenia in the past 6 months.
4. Patient ever attempted to permanently discontinue nilotinib treatment.
5. Known impaired cardiac function including any one of the following:

   * Inability to determine QT interval on ECG
   * Complete left bundle branch block
   * Long QT syndrome or a known family history of long QT syndrome
   * History of or presence of clinically significant ventricular or atrial tachyarrhythmias
   * Clinically significant resting bradycardia
   * QTcF > 480 msec
   * History or clinical signs of myocardial infarction within 1 year prior to study entry
   * History of unstable angina within 1 year prior to study entry
   * Other clinically significant heart disease (e.g. uncontrolled congestive heart failure or uncontrolled hypertension)
6. Severe and/or uncontrolled concurrent medical disease that in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol.
7. History of acute pancreatitis within 1 year prior to study entry or past medical history of chronic pancreatitis.
8. Known presence of a significant congenital or acquired bleeding disorder unrelated to cancer.
9. History of other active malignancy within 5 years prior to study entry except for previous or concomitant basal cell skin cancer, previous cervical carcinoma in situ treated curatively.
10. Patients who have not recovered from prior surgery.
11. Treatment with other investigational agents (defined as not used in accordance with the approved indication) within 4 weeks of Day 1.
12. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection, or gastric bypass surgery).
13. Patients actively receiving therapy with strong CYP3A4 inhibitors and/or inducers, and the treatment cannot be either discontinued or switched to a different medication prior to study entry.
14. Patients actively receiving therapy with herbal medicines that are strong CYP3A4 inhibitors and/or inducers, and the treatment cannot be either discontinued or switched to a different medication prior to study entry. These herbal medicines may include Echinacea, (including E. purpurea, E. angustifolia and E. pallida), Piperine, Artemisinin, St. John's Wort, and Ginkgo.
15. Pregnant or nursing (lactating) women.
16. Women of childbearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for at least 14 days after stopping medication. There is a limited amount of data on pregnancies in patients while attempting treatment-free remission (TFR). If pregnancy is planned during the TFR phase, the patient must be informed of a potential need to re-initiate treatment with nilotinib during pregnancy.

Highly effective contraception methods include:

* Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
* Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
* Male sterilization (at least 6 months prior to screening). The vasectomized male partner should be the sole partner for that subject.
* Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.

In case of use of oral contraception, women should have been stable on the same pill for a minimum of 3 months before starting the study.

Women are considered post-menopausal and not of childbearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (i.e. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks ago.

In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of childbearing potential.

Inclusion Criteria TFR2 stage:

1. Signed informed consent to the TFR2 stage from the patient or from his/her legal representative.
2. Male and female patients 18 years or older.
3. Diagnosis of CP-CML according to the WHO and no previous history of progression to AP/BP CML.
4. First-line treatment with nilotinib for at least 3 calendar years, followed by first TFR attempt.
5. Failed first TFR attempt followed by at least 1 year of nilotinib retreatment before enrollment in TFR2 stage.
6. MR4 or better (BCR-ABL ≤ 0.01% IS) assessed at screening.
7. Patient must meet the following laboratory values at the reinduction screening visit:

   1. Absolute neutrophil count ≥1.0 x 109/L
   2. Platelets ≥75 x 109/L
   3. Hemoglobin (Hgb) ≥ 9 g/dL
   4. Serum creatinine < 1.5 mg/dL
   5. Total bilirubin ≤ 2 x ULN except for patients with Gilbert's syndrome who may only be included if total bilirubin ≤ 3.0 x ULN or direct bilirubin ≤ 1.5 x ULN
   6. AST ≤ 3.0 x ULN
   7. ALT ≤ 3.0 x ULN
   8. Alkaline phosphatase ≤ 2.5 x ULN
   9. Serum lipase ≤ 1.5 x ULN. For serum lipase > ULN - ≤ 1.5 x ULN, value must be considered not clinically significant and not associated with risk factors for acute pancreatitis
   10. Serum levels of potassium, magnesium, total calcium within the normal limits. Correction of electrolytes levels with supplements to fulfil enrolment criteria is allowed.
8. ECOG performance status 0-2.
9. Study subjects must be able to comply with study procedures and follow-up examinations.

Exclusion Criteria TFR2 stage:

1. Patients with known atypical transcript.
2. CML treatment resistant mutation(s) (T315I, E255K/V, Y253H, F359C/V) detected if testing was done in the past (there is no requirement to perform mutation testing at study entry if it was not done in the past).
3. Dose reductions/interruptions due to neutropenia or thrombocytopenia in the past 6 months.
4. Known impaired cardiac function including any one of the following:

   * Inability to determine QT interval on ECG
   * Complete left bundle branch block
   * Long QT syndrome or a known family history of long QT syndrome
   * History of or presence of clinically significant ventricular or atrial tachyarrhythmias
   * Clinically significant resting bradycardia
   * QTcF > 450 msec (male) or > 460 msec (female)
   * History or clinical signs of myocardial infarction within 1 year prior to study entry
   * History of unstable angina within 1 year prior to study entry
   * Other clinically significant heart disease (e.g. uncontrolled congestive heart failure or uncontrolled hypertension)
5. Severe and/or uncontrolled concurrent medical disease that in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol.
6. History of acute pancreatitis within 1 year prior to study entry or past medical history of chronic pancreatitis.
7. Known presence of a significant congenital or acquired bleeding disorder unrelated to cancer.
8. History of other active malignancy within 5 years prior to study entry except for previous or concomitant basal cell skin cancer, previous cervical carcinoma in situ treated curatively.
9. Patients who have not recovered from prior surgery.
10. Treatment with other investigational agents (defined as not used in accordance with the approved indication) within 4 weeks.
11. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection, or gastric bypass surgery).
12. Patients actively receiving therapy with strong CYP3A4 inhibitors and/or inducers, and the treatment cannot be either discontinued or switched to a different medication prior to study entry.
13. Patients actively receiving therapy with herbal medicines that are strong CYP3A4 inhibitors and/or inducers, and the treatment cannot be either discontinued or switched to a different medication prior to study entry. These herbal medicines may include Echinacea, (including E. purpurea, E. angustifolia and E. pallida), Piperine, Artemisinin, St. John's Wort, and Ginkgo.
14. Pregnant or nursing (lactating) women.
15. Women of childbearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for at least 14 days after stopping medication. There is a limited amount of data on pregnancies in patients while attempting treatment-free remission (TFR). If pregnancy is planned during the TFR phase, the patient must be informed of a potential need to re-initiate treatment with nilotinib during pregnancy

Highly effective contraception methods include:

* Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
* Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
* Male sterilization (at least 6 months prior to screening). The vasectomized male partner should be the sole partner for that subject.
* Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.

In case of use of oral contraception, women should have been stable on the same pill for a minimum of 3 months before starting the study.

Women are considered post-menopausal and not of childbearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (i.e. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks ago.

In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of childbearing potential.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Percentage of patients in full treatment-free remission 96 weeks after the start of the consolidation period of TFR1 stage | Baseline of consolidation phase up to 96 weeks of TFR1 stage
  Full Treatment-Free Remission (FTFR) is defined as patients with Major Molecular Response (MMR) or better (i.e. BCR-ABL ≤ 0.1% IS), including those who have totally discontinued treatment during the Treatment-Free Remission (TFR) stage and those who are treated with half the standard dosage.
  Percentage of patients in full treatment-free remission 96 weeks after the start of the consolidation period of TFR1 stage is calculated by dividing the number of patients with no loss of MMR-Major Molecular Response (BCR-ABL ≤ 0.1% (IS) after 96 weeks by the number of patients who entered consolidation of TFR1 stage.
Percentage of patients in treatment-free remission 48 weeks after starting a second attempt at treatment-free remission during TFR2 stage. | Baseline TFR2 phase (week 96 of TFR2 stage) up to week 144 of TFR2 stage
  Treatment-Free Remission (TFR) is defined as patients with MMR or better (i.e. BCR-ABL ≤ 0.1% IS).
  Percentage of patients in TFR 48 weeks after the start of TFR2 phase during TFR2 stage is calculated by dividing the number of patients with no loss of MMR after 48 weeks by the number of patients who entered TFR2 during TFR2 stage.
  Patients who require re-initiation of nilotinib during TFR2 for loss of MMR, and those discontinued from the study will be considered failures.

SECONDARY OUTCOMES:
Percentage of patients who remain in sustained Deep Molecular Response (DMR) at the end of the consolidation period (week 48 TFR1 stage). | Baseline of consolidation period up to 48 weeks (TFR1 stage)
  The percentage of patients in sustained DMR at the end of the consolidation phase (week 48 of TFR1 stage) is calculated by dividing the number of patients in sustained DMR at week 48 of TFR1 stage by the number of patients who entered the consolidation phase of TFR1 stage.
  Sustained DMR: ≥ MR 4.0 (BCR-ABL level ≤0.01% IS) in all of the last 4 BCR-ABL RQ-PCR assessments
Percentage of patients who remain in DMR at the end of the consolidation period (week 48 of TFR1 stage), at 96 weeks and at 144 weeks after the start of the consolidation period of TFR1 stage. | Baseline of consolidation period, week 48, week 96 and week 144 (TFR1 stage)
  The percentage of patients in DMR is calculated by dividing the number of patients in DMR 48, 96 and 144 weeks after the start of the consolidation period in TFR1 stage by the number of patients who entered the consolidation period in TFR1 stage.
  DMR: ≥ MR 4.0 (BCR-ABL level ≤0.01% IS)
Percentage of patients in full treatment-free remission 144 weeks after the start of consolidation ( end of the TFR1 stage.) | Baseline of consolidation period, week 144 of TFR1 stage
  The percentage of patients in full treatment-free remission at week 144 of TFR1 stage is calculated by dividing the number of patients in full treatment-remission at week 144 (TFR1 stage) by the number of patients who entered the consolidation period (TFR1 stage).
  Full Treatment-Free Remission (FTFR) is defined as patients with Major Molecular Response (MMR) or better (i.e. BCR-ABL ≤ 0.1% IS), including those who have totally discontinued treatment during the Treatment-Free Remission (TFR) stage and those who are treated with half the standard dosage.
Percentage of patients with MMR or better at 48, 96, 144 weeks after starting the consolidation period of TFR1 stage | Baseline of consolidation period, week 48, 96 and 144 of TFR1 stage
  The percentage of patients with MMR or better (i.e. BCR-ABL ≤ 0.1% IS) at week 48, 96 and 144 is calculated by dividing the number of patients with MMR at week 48, 96 and 144 of TFR1 stage, regardless of whether they required re-initiation of treatment after the start the study, by the number of patients who entered the consolidation period of TFR1 stage.
Change in BCR-ABL transcript levels after re-start of nilotinib therapy in patients who failed Treatment Free Remission Phase during TFR1 stage. | Restart of nilotinib therapy up to 144 weeks of TFR1 stage
  Change in BCR-ABL levels (International scale), measured by quantitative Polymerase Chain Reaction (PCR), over time after re-start of nilotinib therapy up to 144 weeks in patient who failed Treatment Free Remission Phase in TFR1 stage.
Change in BCR-ABL transcript levels after discontinuation of nilotinib therapy in TFR1 period in TFR1 stage. | Discontinuation of nilotinib therapy in patients in TFR phase up to 144 weeks of TFR1 stage
  Change in BCR-ABL levels (IS), measured by quantitative PCR, over time after discontinuation of nilotinib therapy in TFR1 period up to 144 weeks of TFR1 stage.
Change in BCR-ABL transcript levels during the consolidation period of TFR1 stage. | Baseline of consolidation period up to 48 weeks of TFR1 stage
  Change in BCR-ABL levels (IS), measured by quantitative PCR, over time during the consolidation period to 48 weeks of TFR1 stage.
Full Treatment-Free Survival (FTFS) in TFR1 stage | Baseline of consolidation period up to 144 weeks of TFR1 stage
  FTFS: time from the start of the consolidation period to the earliest occurrence of any of the following events: loss of MMR, reinitiation of treatment due to any cause, progression to accelerated phase (AP)/blast crisis (BC), or death due to any cause.
Treatment-Free Remission rate (TFR rate) after the start of consolidation of TFR1 stage | Baseline of consolidation, week 96 and week 144 of TFR1 stage
  TFR rate at weeks 96 and week 144 of TFR1 stage is calculated by dividing the number of patients with no loss of MMR and no reinitiation of nilotinib after drug discontinuation at weeks 96 and week 144 of TFR1 stage by the number of patients who entered the TFR1 period of TFR1 stage.
Treatment-free survival (TFS) in TFS1 stage | From the start of the TFR phase up to 144 weeks of TFR1 stage.
  TFS: time from the start of the TFR1 period in TFR1 stage to the earliest occurrence of any of the following events: loss of MMR, reinitiation of treatment due to any cause, progression to AP/BC or death due to any cause.
Progression-free survival (PFS) after the start of the consolidation period of TFR1 stage | Baseline of consolidation up to 144 weeks of TFR1 stage
  PFS: time from the start of the consolidation phase of TFR1 stage to progression to AP/BC or death due to any cause, whichever occurs first.
Progression Free Survival (PFS) after the start of TFR1 period of TFR1 stage | From the start of the TFR1 period up to week 144 of TFR1 stage.
  PFS: time from the start of the TFR1 period of TFR1 stage to progression to AP/BC or death due to any cause, whichever occurs first.
Overall Survival (OS) in TFR1 stage | Baseline of consolidation up to 144 weeks of TFR1 stage
  OS: time from start of the study to death due to any cause.
Correlation between clinical and laboratory factors and clinical outcome | Baseline of consolidation phase up to 96 weeks of TFR1 stage
  Statistical correlation between clinical and laboratory correlates at diagnosis (e.g. Sokal Risk scale, demography, type of BCR-ABL transcript) or during previous treatment (e.g. Early Molecular Response=BCR-ABL transcript measured by quantitative PCR <10% after 3 months of first-line treatment with nilotinib at the dose of 300 mg BID) and the achievement of Full Treatment Free Remission and Treatment Free Remission at 96 weeks of TFR1 stage
Number of patients stratified by risk of cardiovascular disease through the Framingham risk score (TFR1 stage) | Baseline of TFR1 stage
  The Framingham risk score will be assessed at the start of TFR1 stage. The Framingham risk score is an algorithm for estimating the combined risk of fatal and non-fatal cardiovascular disease events. The Framingham risk score was developed from the Framingham heart study, and uses sex, age, total cholesterol, HDL, smoking status, and systolic blood pressure for calculating the risk factor: that correlates into a risk category: low, moderate, moderate - high risk, very high. Minimum value=0, maximum value 100. Higher score means a worse outcome, i.e. a higher risk of cardiovascular diseases.
Number of patients stratified by risk of cardiovascular disease through the Systemic Coronary Risk Evaluation (SCORE) (TFR1 stage) | Baseline of TFR1 stage
  The SCORE will be assessed at the start of TFR1 stage. The SCORE is an algorithm for estimating the 10-year risk of fatal cardiovascular disease. The SCORE was developed for use in Europe, and uses sex, age, smoking status, systolic blood pressure, total cholesterol, and total cholesterol/HDL ratio for calculating the risk factor. The SCORE differentiates between high-risk and low-risk countries in Europe and provides different risk charts for the regions.
Percentage of patients eligible for the TFR2 period among patients entering reinduction with asciminib + nilotinib in TFR2 stage | Baseline of TFR2 stage up to week 96 of TFR2 stage
  Eligibility is defined as sustained DMR, defined as no loss of MR4.0 (BCR-ABL level ≤ 0.01% IS) in any BCR-ABL RQ-PCR assessment. The proportion of eligible patients is calculated by dividing the number of eligible patients by the number of patients who entered reinduction of TFR2 stage.
Number of patients with loss of MMR in TFR2 who regain MMR/DMR by the end of the TFR2 stage | Baseline TFR2 phase (week 96 of TFR2 stage) up to week 144 of TFR2 stage
  The proportion of patients who regain MMR/DMR is calculated by dividing the number of patients in MMR/DMR 48 weeks after the start of TFR2 by the number of patients with loss of MMR in TFR2.
  DMR: ≥ MR 4.0 (BCR-ABL level ≤0.01% IS). MMR: BCR-ABL level ≤0.1% IS.
Change in BCR-ABL transcript levels during reinduction of TFR2 stage. | Baseline of TFR2 stage up to week 96 of TFR2 stage
  Change in BCR-ABL levels (IS), measured by quantitative Polymerase Chain Reaction (PCR), over time from baseline of TFR2 stage up to 96 weeks of TFR2 stage.
Change in BCR-ABL transcript levels after restart of nilotinib therapy in patients who failed TFR2 period in TFR2 stage. | Restart of nilotinib therapy up to week 144 of TFR2 stage
  Change in BCR-ABL levels (IS), measured by quantitative PCR, over time after restart of nilotinib therapy in patients who failed TFR2 period up to 144 weeks of TFR2 stage.
Change in BCR-ABL transcript levels after restart of nilotinib therapy in patients who were not eligible for entering the TFR2 period in TFR2 stage. | Restart of nilotinib therapy up to week 144 of TFR2 stage
  Change in BCR-ABL levels (IS), measured by quantitative PCR, over time after restart of nilotinib therapy in patients after restart of nilotinib therapy in patients who were not eligible for entering the TFR2 period up to 144 weeks of TFR2 stage
Change in BCR-ABL transcript levels after discontinuation of asciminib + nilotinib therapy in TFR2 stage. | Discontinuation of asciminib + nilotinib (week 96 of TFR2 stage) up to week 144 of TFR2 stage
  Change in BCR-ABL levels (IS), measured by quantitative PCR, over time after after discontinuation of asciminib + nilotinib therapy up to 144 weeks of TFR2 stage
Treatment-free survival (TFS) in TFR2 stage | From the start of the TFR period of TFR2 stage up to Week 144 of TFR2 stage.
  TFS: time from the start of the TFR period in TFR2 stage to the earliest occurrence of any of the following events: loss of MMR, reinitiation of treatment due to any cause, progression to AP/BC or death due to any cause.
Progression Free Survival (PFS) after the start of TFR2 period of TFR2 stage | From the start of the TFR2 period of TFR2 stage up to week 144 of TFR2 stage.
  PFS: time from the start of the TFR2 period of TFR2 stage to progression to AP/BC or death due to any cause, whichever occurs first.
Overall Survival (OS) in TFR2 stage | Baseline of reinduction period up to week 144 of TFR2 stage
  OS: time from start of the reinduction period (TFR2 stage) to death due to any cause.
Correlation between clinical and laboratory factors and clinical outcome | Baseline of reinduction up to 144 weeks of TFR2 stage
  Statistical correlation between clinical and laboratory correlates at diagnosis (e.g. Sokal Risk scale, demography, type of BCR-ABL transcript) or during previous treatment (e.g. Early Molecular Response=BCR-ABL transcript measured by quantitative PCR <10% after 3 months of first-line treatment with nilotinib at the dose of 300 mg BID) and the achievement of Full Treatment Free Remission, no loss of MMR and no reinitiation of nilotinib therapy at 144 weeks of TFR2 stage
Number of patients stratified by risk of cardiovascular disease through the Framingham risk score (TFR2 stage) | Baseline of TFR2 stage
  The Framingham risk score will be assessed at the start of TFR2 stage. The Framingham risk score is an algorithm for estimating the combined risk of fatal and non-fatal cardiovascular disease events. The Framingham risk score was developed from the Framingham heart study, and uses sex, age, total cholesterol, HDL, smoking status, and systolic blood pressure for calculating the risk factor: that correlates into a risk category: low, moderate, moderate - high risk, very high. Minimum value=0, maximum value 100. Higher score means a worse outcome, i.e. a higher risk of cardiovascular diseases.
Number of patients stratified by risk of cardiovascular disease through the Systemic Coronary Risk Evaluation (SCORE) (TFR2 stage) | Baseline of TFR2 stage
  The SCORE will be assessed at the start of TFR2 stage. The SCORE is an algorithm for estimating the 10-year risk of fatal cardiovascular disease. The SCORE was developed for use in Europe, and uses sex, age, smoking status, systolic blood pressure, total cholesterol, and total cholesterol/HDL ratio for calculating the risk factor. The SCORE differentiates between high-risk and low-risk countries in Europe and provides different risk charts for the regions.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (21):
- Italy (21):
  - Novartis Investigative Site, Bari, BA
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Cagliari, CA
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Catanzaro, CZ
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Pescara, PE
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Reggio Emilia, RE
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Salerno, SA
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Orbassano, TO
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Verona, VR
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Novara

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com